CLINICAL TRIAL: NCT02244073
Title: Individualized Blood Glucose Control in ICU.
Brief Title: Individualized Blood Glucose Control in ICU. The CONTROLING Study. A Double Blinded Multicentric Randomized Study.
Acronym: CONTROLING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data safety monitoring board decision
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013.808; 2013-A00806-39 (Other: ANSM)
Record Dates: First submitted 2014-09-11; First posted 2014-09-18 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness
Keywords: blood glucose target; ICU; insulin; hypoglycemia; hyperglycemia; glycated hemoglobin
MeSH Terms: conditions — Critical Illness; Insulin Resistance; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized blood glucose target (Experimental): Maintain blood glucose in individualized target based on glycated hemoglobin level (A1c); Blood glucose level is maintained bellow 1.59 × A1c - 1.59 (mmol/l).
  Interventions: Drug: Human insulin - Insulin administration to control blood glucose level.
- Conventional blood glucose target (Active Comparator): Maintain blood glucose bellow 10 mmol/l.
  Interventions: Drug: Human insulin - Insulin administration to control blood glucose level.

INTERVENTIONS:
Drug: Human insulin - Insulin administration to control blood glucose level. — On ICU admission, the glycated hemoglobin level (A1c) is measured and insulin IV is possibly administered using a web based nurse driven insulin infusion protocol (https://extranet.chu-lyon.fr/cpg) to maintain blood glucose level below 10 mmol/l. Glycated hemoglobin result triggers patient randomization. Thereafter, during ICU stay, blood glucose level is maintained either below 1.59 × A1c - 1.59 (mmol/l) (Individualized blood glucose target group), or bellow 10 mmol/l (Conventional blood glucose target group).

SUMMARY:
During the last 2 decades, the management of hyperglycemia in critically ill patients has become one of the most discussed topics in the intensive-care field. The initial data suggesting significant benefit from the normalization of blood glucose levels in critically ill patients using intensive intravenous insulin therapy (Van den Berghe G et al. N Engl J Med. 2001) has been tempered by later studies (Finfer S et al. N Engl J Med. 2009). Some studies suggested that strict blood glucose control might benefit in non-diabetic patient and worsen outcomes in diabetics. We hypothesized that an individualized blood glucose target based on glycated hemoglobin measured at ICU admission would improve outcome when compared to a standard care of maintaining blood glucose bellow 10 mmol/l (180 mg/dl). We designed a randomized double blinded study in which Blood glucose control is piloted in both groups by a web-guided protocol that directly gives instruction to nurses (https://extranet.chu-lyon.fr/cpg). The study will enroll 4200 patients in 10 centers. Primary end point is 90 d outcome after randomization.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for INCLUSION in the study if ALL the following criteria are met:

* Patient is 18 year old or older;
* At time of the patient's admission to the ICU the treating ICU specialist expects the patient will require treatment in the ICU that extends beyond the calendar day following the day of admission.

Exclusion Criteria:

* Patients will be EXCLUDED from the study if ONE or MORE of the following criteria are present:

  * Patient or legal surrogate decision maker does not accept the participation to the study;
  * Imminent death (anticipated in less than 48 hours);
  * The treating clinicians are not committed to full supportive care (no resuscitation, no renal replacement therapy limits in dose of vasoactive support);
  * Patient is expected to be eating before the end of the day following admission;
  * Admission in ICU for hypoglycemic encephalopathy or patient at risk for hypoglycaemia ( e.g. known insulin secreting tumour or history of unexplained or recurrent hypoglycaemia or fulminant hepatic failure);
  * If a patient has previously been enrolled in the CONTROLING Study (patients cannot be enrolled in the CONTROLING Study more than once).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2069 (Actual)
Dates: Start 2015-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 90 days after randomization

SECONDARY OUTCOMES:
All-cause mortality | 28 days after randomization and at ICU discharge
Length of intensive care unit stay | 90 days
Need for respiratory support, vasopressor support, dialysis and non-prophylactic antibiotics | during ICU stay (on average 10 days)
incidence and severity of severe hypoglycemia (less than 2.2 mmol/l) | during ICU stay (on average 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Julien BOHE, MD PhD, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (12):
- France (12):
  - Hôpital Nord Franche Comte, Belfort
  - CH de Bourg-en-Bresse, Bourg-en-Bresse
  - Centre Hospitalier de Bourgoin-Jallieu, Bourgoin
  - CH Chartres, Chartres
  - CHU de Clermont Ferrand - Gabriel Montpied, Clermont-Ferrand
  - CHU de Dijon - Complexe Hospitalier du Bocage, Dijon
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nice - Hôpital de l'Archet 1, Nice
  - CH de Polynésie Française, Papeete
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier de Salon de Provence, Salon-de-Provence

REFERENCES:
- [Result] Bohe J, Abidi H, Brunot V, Klich A, Klouche K, Sedillot N, Tchenio X, Quenot JP, Roudaut JB, Mottard N, Thiolliere F, Dellamonica J, Wallet F, Souweine B, Lautrette A, Preiser JC, Timsit JF, Vacheron CH, Ait Hssain A, Maucort-Boulch D; CONTROLe INdividualise de la Glycemie (CONTROLING) Study Group. Individualised versus conventional glucose control in critically-ill patients: the CONTROLING study-a randomized clinical trial. Intensive Care Med. 2021 Nov;47(11):1271-1283. doi: 10.1007/s00134-021-06526-8. Epub 2021 Sep 29. PMID 34590159
- See also: Related Info — https://extranet.chu-lyon.fr/